CLINICAL TRIAL: NCT01854190
Title: Evaluation of Obstructive Sleep Apnea and Endothelial Function in Resistant Hypertension Patients
Brief Title: Obstructive Sleep Apnea and Endothelial Function in Patients With Resistant Hypertension
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Antonio Felipe Sanjuliani, Doctor / Professor, Rio de Janeiro State University
Other Study IDs: CLINEX 02
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-02

CONDITIONS: Obstructive Sleep Apnea; Secondary Hypertension
Keywords: Obstructive sleep apnea; Resistent hypertension; Endothelial function; Blood pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Resistant hypertension: Patients with uncontrolled blood pressure despite 3 medications, including diuretic.
  Endothelial function assessed by peripheral arterial tonometry (PAT) by EndoPAT and the OSA diagnosis also through PAT, using the portable device WatchPAT.
  Interventions: Device: WatchPAT
- Controlled hypertension: Patients with controlled blood pressure by medications. These drugs are the same used in both groups.
  Interventions: Device: WatchPAT

INTERVENTIONS:
Device: WatchPAT — BP was measured by oscillometric method on automatic device. Endothelial function was assessed by peripheral arterial tonometry (PAT) by EndoPAT2000® and the OSA diagnosis also through PAT, using the portable device WatchPAT200®. Anthropometric evaluation was performed through measurements of waist, hip and neck circumference, body mass index, waist to height ratio (WHtR), and body composition assessed by bioelectrical impedance.
  Other Names: WatchPAT 200 - Itamar Medical; EndoPAT 2000 - Itamar Medical; Omron 742INT

SUMMARY:
The purpose of this study is to determine the prevalence of obstructive sleep apnea and associate it with the endothelial function behavior in patients with resistant hypertension. Two groups will be evaluate, one presenting uncontrolled high blood pressure, and other, with controlled blood pressure by drugs.

DETAILED DESCRIPTION:
Introduction: Obstructive sleep apnea (OSA) is considered an independent risk factor for cardiovascular disease. There is evidence that individuals with OSA may have increased inflammatory mediators, changes in the metabolic profile, increased sympathetic activity with consequent elevation of blood pressure (BP) and endothelial dysfunction. Resistant hypertension (RH) is defined as uncontrolled blood pressure (BP ≥ 140/90mmHg) despite the current use of three hypotensive drugs at full doses, including a diuretic, or the need for >3 medications to control BP. OSA has been reported as the most common secondary cause of high blood pressure maintenance.

Objective: To determine the prevalence of OSA and associate it with the endothelial function behavior in patients with resistant hypertension comparing to those with BP controlled by medication.

Methods: A cross-sectional study involving 40 hypertensive patients (20 with resistant hypertension and 20 with controlled BP), irrespective of race or gender, with ages between 18 and 75 years. BP was measured by oscillometric method on automatic device. Endothelial function was assessed by peripheral arterial tonometry (PAT) by EndoPAT2000® and the OSA diagnosis also through PAT, using the portable device WatchPAT200®. Anthropometric evaluation was performed through measurements of waist, hip and neck circumference, body mass index, waist to height ratio (WHtR), and body composition assessed by bioelectrical impedance. Statistical analyzes were performed by GraphPad Prism software.

ELIGIBILITY:
Inclusion Criteria:

* ages between 18 and 75 years
* previous hypertension diagnosis

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients, from the Hypertension Clinic of UERJ
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive sleep apnea | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F Sanjuliani, MD, ScD, Principal Investigator — Rio de Janeiro State University - Brazil
Locations (1):
- Pedro Ernesto University Hospital, Rio de Janeiro, Rio de Janeiro, Brazil